CLINICAL TRIAL: NCT01523431
Title: Influence of Individual Dosage Selection of Irinotecan (CPT-11) Based on UGT1A1 Genotype on Clinical Outcomes and Pharmacokinetics in Chinese Patients With Metastatic Colorectal Cancer
Brief Title: Individual Dosage Selection of Irinotecan (CPT-11) Based on UGT1A1 Genotype in Metastatic Colorectal Cancer Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other)
Responsible Party: Principal Investigator, Xu jianming, Director of Department of GI Cancer, The Affiliated Hospital of the Chinese Academy of Military Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCRC-307PLAH-XJM
Record Dates: First submitted 2012-01-19; First posted 2012-02-01 (Estimated); Last update posted 2017-03-30 (Actual); Status verified 2017-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Colorectal cancer; Irinotecan; UGT1A1 genotype; Neutropenia; diarrhea; response; pharmacokinetic
MeSH Terms: conditions — Colorectal Neoplasms; Neutropenia; Diarrhea | interventions — Irinotecan; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard FOLFIRI for wild/hetero UGT1A1 (Active Comparator): Irinotecan Injection [Camptosar] (CPT-11) 180 mg/m2, day 1; Leucovorin (LV) 400mg/m2, day 1; 5-fluorouracil (5-FU) 400mg/m2, day 1, 5-fluorouracil (5-FU) 2400mg/m2, day 1; Repeat every two weeks.
  Interventions: Drug: Irinotecan Injection [Camptosar]; Drug: 5-fluorouracil; Drug: Leucovorin
- Reduced Dose of CPT-11 for homo UGT1A1 (Experimental): Irinotecan Injection [Camptosar] (CPT-11) 90 mg/m2, day 1; Leucovorin (LV) 400mg/m2, day 1; 5-fluorouracil (5-FU) 400mg/m2, day 1, 5-fluorouracil (5-FU) 2400mg/m2, day 1; Repeat every two weeks.
  Interventions: Drug: Irinotecan Injection [Camptosar]; Drug: 5-fluorouracil; Drug: Leucovorin
- Standard FOLFIRI for homo UGT1A1 (Active Comparator): Irinotecan Injection [Camptosar] (CPT-11) 180 mg/m2, day 1; Leucovorin (LV) 400mg/m2, day 1; 5-fluorouracil (5-FU) 400mg/m2, day 1, 5-fluorouracil (5-FU) 2400mg/m2, day 1; Repeat every two weeks.
  Interventions: Drug: Irinotecan Injection [Camptosar]; Drug: 5-fluorouracil; Drug: Leucovorin

INTERVENTIONS:
Drug: Irinotecan Injection [Camptosar] — CPT-11 will be administered according to UGT1A1 genotypes. Patients with UGT1A1 *1/*1 or heterozygous UGT1A1*1/*28 or *1/*6 will receive standard dose of CPT-11. Patients with homozygous UGT1A1*28/*28, *6/*6 or *28/*6, will be randomized in a 1:1 ratio to receive standard dose of CPT-11 or 50% reduced dose of CPT-11.
  Other Names: CPT-11; FOLFIRI regimen
Drug: 5-fluorouracil — The 5-FU dosage will remain the standard.
  Other Names: 5-FU; FOLFIRI regimen
Drug: Leucovorin — The LV dosage will remain the standard.
  Other Names: LV; FOLFIRI regimen

SUMMARY:
The purpose of this study is to investigate the influence of dose selection of CPT-11 on toxicity, response and pharmacokinetics according to UGT1A1 genotype in colorectal cancer patients.

DETAILED DESCRIPTION:
Genetic polymorphisms of UGTs result in reduced enzyme activity and increased toxicity. UGT1A1*28 and UGT1A1*6 are reported to increase CPT-11-related toxicity in Asian patients. Moreover, the area under concentration curve (AUC) ratio of SN-38G to SN-38 is decreased in Asian patients having UGT1A1 *28 or UGT1A1*6. This implicated that the current standard dose of CPT-11 would be overdosing for homozygous UGT1A1*28/*28, *6/*6 or *28/*6 patients.

The study is designed to investigate the role of prospectively dose reduction of CPT-11 in toxicity, tumor response and pharmacokinetics for homozygous UGT1A1 patients, and compare these parameters to standard dose of CPT-11 for wild-type, heterozygous or homozygous UGT1A1 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed colorectal cancer patients who received no prior chemotherapy or failed to 1st line treatments
2. At least one measurable lesion by Response Evaluation Criteria in Solid Tumors (RECIST) criteria
3. Aged 18 years or older
4. ECOG performance status of ≤ 2.
5. Anticipated life expectancy of ≥ 3 months.
6. UGT1A1 genotype tested. Categorized into Wild (UGT1A1*1/*1), Hetero (UGT1A1*1/ *28, UGT1A1*1/ *6), and Homo (UGT1A1*28/*28, UGT1A1*6/*6, UGT1A1*28/*6).
7. Adequate organ function, including bone marrow, kidney and liver.

   * ANC ≥ 1.5×109/L and hemoglobin ≥ 9g/dL and platelet count ≥ 100×109/L
   * Serum total bilirubin ≤ 1.5 x ULN, alkaline phosphatase ≤ 2.5 x ULN, Serum ALT and AST ≤ 2.5 x ULN (Serum ALT and AST ≤ 5 x ULN, if liver metastases are present)
   * Serum creatinine ≤ 1.5 x ULN or CLcr > 60 ml/min
8. Written informed consent can be obtained prior to their participation in the trial.

Exclusion Criteria:

1. Pregnant or breast feeding women.
2. Subjects who have previously received CPT-11 treatment.
3. Serious concurrent complication, severe active infection.
4. Subjects with chronic diarrhea, acute or sub acute Intestinal obstruction.
5. Subjects with uncontrolled CNS metastasis or epilepsia or severe psychiatric disorders.
6. Subjects who are regarded to be unsuitable for this trial by the investigator.
7. Subjects who are participating in other clinical trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 583 (Actual)
Dates: Start 2012-03-08 (Actual); Primary Completion 2015-11-23 (Actual); Study Completion 2016-04-27 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicity, especially neutropenia and diarrhea | From the beginning of treatment to the whole treatment period, an expected average of 6-8 months.
  Association between UGT1A1 polymorphism, CPT-11 dosage and incidence of toxicity, especially neutropenia and diarrhea.

SECONDARY OUTCOMES:
Response rate | Every 6 weeks, an expected average of 6-8 months.
  Association between UGT1A1 polymorphism, CPT-11 dosage and tumor response.
Progression-free survival (PFS) | An expected average of 6-8 months.
  Association between UGT1A1 polymorphism, CPT-11 dosage and PFS. PFS is defined as the length of time from randomise to disease progression or to death from any cause other than progression.
Pharmacokinetics of irinotecan and its metabolites, SN-38 and SN-38G. | The first treatment cycle.
  Association between UGT1A1 polymorphism, CPT-11 dosage and pharmacokinetics of irinotecan. Plasma concentration of irinotecan and its metabolites, SN-38 and SN-38G are determined using high-performance liquid chromatography-tandem mass spectrometry method (HPLC-MS/MS).

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Ming Xu, M.D., Principal Investigator — Affiliated Hospital, Academy of Military Medical Sciences
Locations (1):
- Affiliated Hospital Cancer Center, Academy of Military Medical Sciences (307 Hospital of PLA), Beijing, Beijing Municipality, China